CLINICAL TRIAL: NCT03197740
Title: A Multinational, Multi-center, Randomized, Double-blind, Active Comparator, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Donepezil Transdermal Patch in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icure Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPI-003
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- aricept Tab 5mg (Active Comparator)
  Interventions: Drug: aricept Tab
- donepezil patch 25cm2 (Experimental)
  Interventions: Drug: Donepezil patch
- aricept Tab 10mg (Active Comparator)
  Interventions: Drug: aricept Tab
- donepezil patch 50cm2 (Experimental)
  Interventions: Drug: Donepezil patch

INTERVENTIONS:
Drug: Donepezil patch — Treatment
  Arms: donepezil patch 25cm2; donepezil patch 50cm2
Drug: aricept Tab — Comparator
  Arms: aricept Tab 10mg; aricept Tab 5mg

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of donepezil transdermal patch in patients with mild to moderate Alzheimer's disease.

The primary objective is to demonstrate the non-inferiority of the test drug, IPI-301 (donepezil transdermal patch), to the comparator, Aricept tablet, after 24 weeks of treatment in patients with mild to moderate Alzheimer's disease in terms of improvement in cognitive function as assessed by the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog) and in terms of global assessment as assessed by Clinician's Interview Based Impression of Change plus Caregiver Input (CIBIC-plus).

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥50 to ≤85 as of the date of informed consent
2. Clinical diagnosis of probable Alzheimer's disease according to Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV) and National Institute of Neurological and Communicative Disorders and Strokes; Alzheimer's disease and Related Disorders Association (NINCDS-ADRDA)
3. Mini Mental Status Examination (MMSE) score ≥10 to ≤26 at screening
4. Global Clinical Dementia Rating (CDR) score 0.5, 1 or 2 at screening
5. Capable of performing procedures for cognitive and other tests
6. Subject who meets any of the following as of the date of informed consent

   * No past treatment with donepezil (naïve patient)
   * Ongoing treatment with donepezil 10mg/day for the past 3 months
   * Ongoing treatment with donepezil 5mg/day for the past 3 months
7. The subject or his/her representative must voluntarily decide to participate in the study and provide written informed consent.
8. The subject must have a reliable caregiver who regularly contacts the subject and is available to accompany the subject for on-site visits. (Note: A caregiver is defined as someone who has regular contact with the subject [i.e., an average of approximately 10 or more hours per week], must be able to oversee subject's compliance with the study treatment and to report on the patient's status and must be able to accompany the subject to all study visits.)

Exclusion Criteria:

1. Possible, probable, or definite vascular dementia according to National Institute of Neurological Disorders and Stroke/Association Internationale pur la Recherche et I'Enseignement en Neurosciences (NINDS-AIREN)
2. History and/or evidence (computed tomography [CT] or magnetic resonance imaging [MRI] findings obtained within the past 12 months or at screening) of other central nervous system (CNS) disorders (cerebrovascular disease, structural or developmental anomaly, epilepsy, or communicable, degenerative, or infectious/demyelinating CNS conditions) as a cause of dementia Note: >3 lacunar infarcts over 10 mm each, or severe white matter disease equaling a rating of 3 on the age-related white matter changes (ARWMC scale) should be excluded in the study.
3. Illiteracy
4. Treatment with other anti-dementia drugs (galantamine, memantine, rivastigmine, tacrine), except donepezil, within the past 3 months from the date of informed consent
5. Treatment with any of the following drugs within the past 2 weeks from the date of informed consent

   * CNS stimulants: methylphenidate, modafinil, pemoline, atomoxetine
   * Typical antipsychotics: bromperidol, chlorpromazine, haloperidol
   * Anticholinergics: atropine, glycopyrrolate, scopolamine, homatropine, ipratropium (short term [within 3 days] use of anticholinergics for the purpose of antispasmodic action on the digestive system is permitted.)
6. Abnormal blood test findings as follows at the screening test:

   * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≥2.5 x upper limit of normal
   * A serum creatinine level of ≥1.5 × ULN for the reference laboratory, or a calculated creatinine clearance by the Cockcroft-Gault equation of ≤50mL/min
7. Clinically significant abnormal vitamin B12, syphilis serology, or thyroid stimulating hormone (TSH) test findings considered to contribute to the severity of dementia or to be attributable to dementia

   Note:
   1. Clinically significant untreated B12 should be excluded in the study. Subjects are eligible if B12 deficiency is stable after the treatment.
   2. If the subject has tested False positive for syphilis test, based on the investigator's judgment, further test can be performed to get the final result.
   3. TSH >10mIU/L should be excluded in the study.
8. Diagnosis of serious mental disease based on DSM-5 criteria, including depressive disorder,, schizophrenia, alcoholism, drug dependency, etc.
9. Parkinson's disease or parkinsonian syndrome
10. Clinically significant electrocardiogram (ECG) abnormalities at screening (heart rate <50 beats/min, atrial and ventricular conduction disorders such as 2nd degree atrioventricular block, QTc interval >480ms)
11. History of unstable angina pectoris, myocardial infarction, transient ischemic attack, or coronary intervention including coronary bypass within the past 6 months from the date of informed consent
12. History of severe traumatic head injury with loss of consciousness within the past 6 months from the date of informed consent
13. Asthma or obstructive pulmonary disease requiring medication
14. Gastrointestinal disorders that may affect the absorption, distribution, and metabolism of the study drug (e.g., inflammatory bowel disease, gastric or duodenal ulcer, hepatic disease)
15. Uncontrolled diabetes mellitus (defined as HbA1c>9.0%)
16. Administration of other investigational products within 3 months prior to treatment with the investigational product (Day 0)
17. Hypersensitivity reactions to donepezil HCl, piperidine derivatives, or any of the components of the study drug
18. Pregnant or lactating woman or woman of childbearing potential who does not agree to use an effective method of contraception.

    : Recommended effective methods of birth control include diaphragm plus spermicide or male condom plus spermicide, oral contraceptive in combination with a second method, contraceptive implant, injectable contraceptive, indwelling intrauterine device, sexual abstinence, and vasectomized partners. The subject/investigator can discuss any other best method that suits the subject.
19. Hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
20. Human immunodeficiency virus (HIV) positive or Acquired Immune Deficiency Syndrome (AIDs)
21. History of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured, and cervical carcinoma in situ). Cancer survivors not on maintenance therapy that had no malignant disease history within the past 5 years could be recruited.
22. Individual considered by the investigator to be ineligible for study participation for other reasons, including having a condition that may affect the assessment of study results

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
ADAS-cog | week 24
  Change at Week 24 of treatment with the study drug from baseline (0d) in ADAS-cog scores

SECONDARY OUTCOMES:
CIBIC-plus | week 24
  CIBIC-plus score at the end of treatment (Week 24)

CONTACTS AND LOCATIONS:
Locations (1):
- 46 Sites including Konkuk University Medical Center, Seoul, South Korea